CLINICAL TRIAL: NCT00937690
Title: Pilot Study of Infrared Imaging of Cutaneous Melanoma
Acronym: MEL49
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Sponsor
Other Study IDs: 13564
Record Dates: First submitted 2009-06-01; First posted 2009-07-13 (Estimated); Last update posted 2014-12-23 (Estimated); Status verified 2014-12

CONDITIONS: Melanoma
Keywords: melanoma; cutaneous; imaging
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- infrared imaging of cutaneous lesions: patients and volunteers with cutaneous lesions, with and without clinically detectable melanoma, and with one or more palpable cutaneous lesions

SUMMARY:
Design: this is a pilot study of infrared imaging of cutaneous lesions in patients and volunteers with and without clinically detectable melanoma, and with one or more palpable cutaneous lesions eligible for this imaging study. Participants will be evaluated with infrared camera imaging at cutaneous sites with known melanoma deposits, suspected melanoma deposits that are to be biopsied, or at cutaneous sites with other lesions, including other skin cancers, benign inflammatory lesions, benign neoplastic lesions (lipomas, epidermal cysts, dermatofibromas, scar, healing wound, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Patients or volunteers with or without a history of melanoma.
* One or more palpable skin or subcutaneous lesions for which at least one of the following is true:

  * A tissue diagnosis has been made for the lesion(s) in question, by prior cytologic or histologic evaluation (Category A1).
  * A tissue diagnosis will be obtained for the lesion(s) in question by cytologic or histologic evaluation (Category A2).
  * A tissue diagnosis is not available, but a clinical diagnosis of melanoma or benign lesion is available with a high degree of confidence. Examples are hemangiomas, skin tags, seborrheic keratoses, dermatofibromas, lipomas, or growing pigmented skin lesions that are comparable to other cutaneous metastases of melanoma in the same patient (Category B).
* All patients must have the ability and willingness to give informed consent and must be age 18 years or older at the time of study entry.

Exclusion Criteria:

* Known or suspected allergy to the adhesive skin markers or water-soluble ink used for the labeling of lesions.
* Very fragile skin that may be susceptible to injury from adhesive markers.
* Patients in whom there is a medical contraindication or potential problem in complying with the requirements of the protocol, in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients and volunteers over the age of 18 with palpable cutaneous skin lesions. Patients of all races and ethnic backgrounds are eligible. Efforts will be made to include pigmented and non-pigmented lesions in participants with a range of skin colors, including skin-colored papules in African-American and Hispanic patients when available.
Sampling Method: Non-Probability Sample
Enrollment: 74 (Actual)
Dates: Start 2008-03; Primary Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
preliminary estimate sensitivity of infrared imaging in detecting melanoma metastasis as function of lesion diameter | one day - 24 hours

SECONDARY OUTCOMES:
to obtain preliminary estimate of specificity of infrared imaging for detection of melanoma metastasis | one day-24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Craig L Slingluff, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States